CLINICAL TRIAL: NCT01301300
Title: Demonstration of Central Line Hub Contamination Reduction Using a Novel Capping Device
Brief Title: Evaluating Central Line Hub Contamination Using a Novel Capping Device
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Endeavor Health (Other)
Responsible Party: Lance R Peterson, Associate Hospital Epidemiologist, NorthShore University Health System
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EH10-125
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Catheter-related Bloodstream Infection Due to Central Venous Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glenbrook Hospital (Active Comparator): Immediate implementation of the disinfecting cap, no baseline contamination assessment, historical infection data only.
  Interventions: Device: Disinfecting Cap
- Evanston, Highland Park, Skokie Hospitals (Active Comparator): Phase 1: Assess baseline contamination rate for patients with PICC catheters for 3-12 months.
  Phase 2: Implement intervention. Assess contamination 3-12 months. Phase 3: (optional): Remove cap asses contamination rate (3-6 months)
  Interventions: Device: Disinfecting Cap

INTERVENTIONS:
Device: Disinfecting Cap — Replace standard practice with using the disinfecting cap
  Other Names: SwabCap SC003 2000

SUMMARY:
Excelsior Medical has developed SwabCap™, a luer access valve disinfection cap. The SwabCap™ provides passive disinfection of valve top and threads without activating the luer access valve. This product promotes technique standardization and compliance in cleansing of the luer access valve prior to access. It acts as a physical barrier from touch and airborne contamination for up to 96 hours. This product has been endorsed and will be adopted for use at NorthShore University HealthSystem as a quality improvement initiative. This research study protocol is designed to confirm the anticipated benefit of this change in practice at NorthShore during the planned implementation and use.

If the product performs as it has been designed to, the baseline rate of hub and subsequently intraluminal contamination will be diminished, thereby protecting patients with central lines from bloodstream infections due to contaminated hubs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with peripherally inserted central catheters (PICC) inserted during their index hospitalization plus 5 or more consecutive PICC line days were consented and enrolled.

Exclusion Criteria:

* Minors and adult inpatients without PICCs or with PICCs for < 5 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative contamination of intraluminal fluid from central venous catheters (discard) as measured in CFU/ml | Throughout the study with enrolled subjects (The catheter must have been in place for a period of 5 or more days before the first sample is taken.)
  For the research project, we will monitor the colonization of access port colonization in routine as well as SwabCap™ cared for lines as follows:
  Specimen sampling will be done by obtaining one specimen of 1.0 mL of aspirate will be withdrawn from each unused catheter lumen during first morning rounds in a separate syringe; then placed in a epdiatric Isolator tube.

SECONDARY OUTCOMES:
Central line associated bloodstream infections | Throughout the study and from historical data
  Central line-associated bloodstream infections (CLABSI) as defined by the National Healthcare Safety Network (NHSN) of all patients throughout 4 hospitals in 2009-2011.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - NorthShore: Evanston Hospital, Evanston, Illinois
  - NorthShore: Glenbrook Hospital, Glenview, Illinois
  - NorthShore: Highland Park Hospital, Highland Park, Illinois
  - NorthShore: Skokie Hospital, Skokie, Illinois